CLINICAL TRIAL: NCT04718441
Title: Contrast Ultrasound for Pediatric Trauma - Comparative Evaluation (CAPTURE Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Mooney (Other)
Responsible Party: Sponsor-Investigator, David Mooney, Director Trauma Program, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P00035263
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Abdominal Injury
Keywords: Solid Organ Injury
MeSH Terms: conditions — Abdominal Injuries | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Study Participants (Experimental): All subjects will have an abdominal non-contrast ultrasound performed. Lumason will then be administered at a dose of 0.03mL/kg up to a maximum dose of 2.4mL and a contrast-enhanced ultrasound will be performed. The dose will be given twice, for a total maximum dose per subject of 4.8mL
  Interventions: Drug: Lumason

INTERVENTIONS:
Drug: Lumason — Lumason will be administered at a dose of 0.03 mL/kg up to a maximum dose of 2.4mL injected into a peripheral intravenous catheter. An abdominal contrast enhanced ultrasound will be performed to look for solid organ injury. The will be given twice during the intervention, for a total maximum dose per subject of 4.8mL.
  Other Names: SonoVue

SUMMARY:
This multicenter study aims to evaluate the accuracy of contrast-enhanced ultrasound (CEUS) in diagnosing abdominal solid organ injuries in pediatric patients. Up to 130 subjects will complete the study across approximately 5-10 sites in the US, with up to 30 patients in the training phase (3 per site) and 100 patients in the treatment phase of the study. All subjects will have had a CT scan as part of standard of care, confirming at least one solid organ abdominal injury. The study procedure will occur within 48 hours from time of injury. All subjects will have an abdominal ultrasound without contrast, followed by a contrast-enhanced ultrasound using the contrast agent Lumason. Ultrasound and contrast-enhanced ultrasound results will be compared to the CT scan results. The CT and ultrasound scans will be read locally and will undergo central review.

DETAILED DESCRIPTION:
This is an interventional study which proposes to evaluate the accuracy of contrast-enhanced ultrasound (CEUS) in diagnosing abdominal solid organ injuries in pediatric trauma patients. Up to 130 subjects will be enrolled across approximately 5 to 10 sites in the US. Each site, including the coordinating center, will undergo the training phase; each site will enroll 3 participants in this phase successfully prior to entering the treatment phase. All subjects will have had a Computerized Tomography (CT) scan as part of standard of care, confirming at least one solid organ abdominal injury. All subjects will have an abdominal ultrasound without contrast, followed by a contrast-enhanced ultrasound using the contrast agent Lumason. Ultrasound and contrast-enhanced ultrasound results will be compared to the CT scan results. The study procedures will take place within 48 hours of injury. At conclusion of enrollment of all subjects a centralized review of CT vs. CEUS will occur to compare to real-time readings.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodynamically stable, as determined by the trauma team
2. Age 8 through 18 years (inclusive)
3. Interpretable CT of the abdomen and pelvis that demonstrates at least one solid organ injury among the liver, spleen, pancreas, and kidneys
4. Plan for observation or admission to the hospital
5. Candidate for abdominal ultrasound based on body habitus, as determined by the investigator
6. Glasgow Coma Score of 15
7. Able to complete the study procedures within 48 hours of injury

Exclusion Criteria:

1. Known cardiac abnormality
2. Pulmonary Hypertension
3. Known sensitivity to any Lumason components - including sulfur hexafluoride, polyethylene glycol 4000, distearoylphosphatidylcholine (DSPC), dipalmitoylphosphatidylglycerol sodium (DPPG-Na), or palmitic acid
4. Unable to be rolled onto side to allow lateral ultrasound windows if necessary
5. Unable to assent or consent
6. Pregnant
7. Lactating
8. CT images not available for transmission to central image repository

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Overall CEUS/CT Concordance for all study participants | At the time the CEUS is performed, within 48 hours of injury
  A patient is classified as having a "concordant" assessment if each organ identified by CT with injuries is exactly identified by CEUS, regardless of injury grade, by the local study site reviewer. Otherwise, a patient is classified as having a "discordant" assessment.

SECONDARY OUTCOMES:
Organ-specific CEUS/CT Concordance | At the time the CEUS is performed, within 48 hours of injury
  For each organ, a patient's organ is classified as having a "concordant" assessment if the presence or absence of an injury as identified by CT is exactly identified by CEUS. Otherwise, a patient is classified as having a "discordant" assessment.
Grade-specific Overall CEUS/CT Concordance | At the time the CEUS is performed, within 48 hours of injury
  A patient is classified as having a "concordant" assessment if each organ identified by CT with injuries is exactly identified by CEUS, AND within 1 grade of the injury as identified by CT. Otherwise, a patient is classified as having a "discordant" assessment.
Peritoneal Fluid CEUS/CT Concordance | At the time the CEUS is performed, within 48 hours of injury.
  A patient is classified as having a "concordant" assessment if the absence or presence of peritoneal fluid identified by CT is also exactly identified by CEUS. Otherwise, a patient is classified as having a "discordant" assessment.
Real-time/Centralized CEUS Concordance | At the time the CEUS is performed, within 48 hours of injury.
  A patient is classified as having a "concordant" assessment if the absence or presence of injury for each organ identified by 'real-time' CEUS with injuries is also exactly identified by centralized interpretation of CEUS images.

CONTACTS AND LOCATIONS:
Overall Officials: David Mooney, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (5):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah